CLINICAL TRIAL: NCT00713869
Title: Evaluation of the Affects of an Oocyte Freezing and Thawing Technique in Patients Undergoing In-vitro Fertilization (IVF)
Brief Title: Oocyte Cryopreservation: Evaluation of an Oocyte Freezing and Thawing Technique
Acronym: Slow-freeze
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: West Coast Fertility Centers (Other)
Responsible Party: David G. Diaz MD, West Coast Fertility Centers
Other Study IDs: 20052092
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Infertility
Keywords: Oocyte cryopreservation; Slow freeze
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients between the ages of 21 and 35 undergoing in-vitro fertilization will be included in this study.
- 2: Recipients using only frozen donor eggs

SUMMARY:
Over the past several decades, considerable effort has been expended toward the successful cryopreservation of various human cells. While attempts at cryopreservation have been directed at different tissue types, one of the most vigorously pursued targets has been reproductive tissue. Historically, cryopreservation of human sperm has existed for several decades. The earliest reports of pregnancies (Trounson et al., 1983) and births (Zeilmaker et al., 1984) from the cryopreservation of human embryos occurred in the early 1980s. Presently, the freezing and storage of human embryos following in vitro fertilization (IVF) is standard practice at most fertility clinics. In 2003, the CDC Assisted Reproductive Technology success rates report stated that 4,246 live births occurred out of 17,517 non-donor frozen embryo cycles. . Because the human egg is a relatively voluminous cell with abundant cytoplasm, crystallization at the time of freezing may result in damage to the organelles. Secondly, a mature metaphase II oocyte contains a fragile spindle apparatus involved in cleavage.

The purpose of this research study is to evaluate a method of freezing and thawing oocytes. This evaluation will be made by comparing the survival rates and rates of fertilization, cleavage and embryo quality of fresh oocytes and frozen-thawed oocytes which will be inseminated during the IVF (in vitro fertilization) treatment cycle. In addition, the same comparisons will be made between frozen oocytes from infertile women and those of egg donors. You are being asked to be in this study because you are currently undergoing in vitro fertilization.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into this study, each subject must satisfy the following criteria:

1. Infertile woman wishing to conceive and whose physician has recommended that she undergo IVF.
2. Participants must be aged 21 to 35 years
3. Body mass index (BMI) < 38.
4. Serum results for cycle day 3 FSH <10 mIU/ml.
5. Must have male partner whose semen analysis meets the clinic criteria for ICSI. Use of donor sperm is also acceptable.
6. Be willing and able to comply with the protocol for the duration of the study.
7. Have voluntarily provided written informed consent under WIRB, prior to any study-related procedure that is not part of normal medical care, with the understanding that the subjects may withdraw consent before they start Lupron without prejudice to their future medical care.

Exclusion Criteria:

A patient may NOT be entered into the study if she presents with ANY of the following criteria:

1. Clinically significant systemic disease.
2. Known endometriosis Grade III - IV (ASRM classification).
3. Any previous cycle indicating a low response to gonadotropin stimulation (defined as retrieval of < 10 eggs at retrieval)
4. Three or more previous ART cycles without a clinical pregnancy
5. Abnormal, undiagnosed, gynecological bleeding.
6. Previous ovarian surgery
7. Known allergy or hypersensitivity to recombinant gonadotropin preparations or any other study-related medications.
8. Known current substance abuse.
9. Simultaneous participation in another clinical trial.
10. Current smoker.
11. An extrauterine pregnancy within the last 3 months before OCP treatment commences.
12. Previous participation in similar study at different centers.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertility patient
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-11 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Freeze / thaw survival rates. Fertilization rates. Cleavage rates. Embryo quality measured by pronuclear and day 2 morphology. | When oocyte thawed initiate.

CONTACTS AND LOCATIONS:
Overall Officials: David G. Diaz, MD, Principal Investigator — West Coast Fertility Centers
Locations (1):
- West Coast Fertility Centers, Fountain Valley, California, United States